# **RUST - Rusfri Uten Tannverk**

Målsetninger: Denne feasibility/pilotstudiens primære målsetning er å undersøke gjennomføringsgraden av tannbehandling i løpet av oppholdet ved UNN Russeksjon Narvik. Med andre ord: Hvor mange gjennomfører gratis tannbehandling hvis de får tilbud om det? Den sekundære målsetningen er å kartlegge hvilke assosiasjoner som øker sannsynlighet for gjennomføring. Disse assosiasjonene skal brukes til å modellere risiko for frafall fra tannbehandling.

I tillegg vil vi undersøke om parallell tannbehandling har innvirkning på utbytte av rusbehandlingen, eller om det kan virke forstyrrende for gjennomføring.

Metodologi: RUST er en intervensjonsstudie uten kontrollgruppe der et tilbud om tannbehandling implementeres parallelt med rus- og avhengighetsbehandling. I studien vil vi inkludere 40-50 pasienter som legges inn ved UNN Russeksjon Narvik i 2021. Deltakerne følges under behandlingstiden, forventet varighet er omkring 12 uker for den enkelte. Alle som inkluderes får tannbehandling i løpet av behandlingsoppholdet. Informasjon om deltakernes rusbruk og tann/munnhelse samles inn med spørreskjema før, under og etter studien. For primær målsetning (gjennomføringsgrad av tannbehandling) vil det gjøres deskriptive statistiske analyser av gjennomføringsgrad for å etablerer den prosentvise fordelingen. For sekundær målsetning (assosiasjoner som øker sannsynlighet for gjennomføringsgrad) vil det lages en klassifiseringsmodell som kan oppgi sannsynlighet for frafall, basert på informasjon fra journal og spørreskjema ved inklusjon. Enkle modeller vil først bli benyttet (f.eks. basert på logistisk regresjon eller naive bayes) for å gi et grunnlag for å vurdere potensialet til framgangsmåten.

Hvorvidt tannbehandling kan virke positivt eller negativt for rusbehandling vil utforskes ved hjelp av spørreskjema og samtaler med deltakere.

**Endepunkter:** Primært endepunkt er andel pasienter som gjennomfører tannbehandling i løpet av innleggelsen. Tannlegen vil definere om behandlingen ble gjennomført på tilstrekkelig vis ut fra planlagt tannbehandling ved første konsultasjon.

Sekundært endepunkt, utvikle en klassifiseringsmodell for hvilke faktorer som påvirker sannsynlighet for gjennomføring av tannbehandling. Klassifiseringsmodellen skal vurderes på testegenskaper som sensitivitet, spesifisitet, likelihood ratio og område under receiver operating characteristics curve (ROC kurve). For å kunne sies å være nyttig må dette verktøyet være beviselig bedre enn et overslag basert på hvor mange som gjennomfører på helt generell basis (etablert i målsetning 1).

Betydning: Resultatene av studien vil være med på å avklare om det vil være meningsfullt å implementere gratis tannbehandling som et ordinært tilbud i klinisk sammenheng. Høy andel av gjennomføring vil også gjøre det mulig å studere behandlingseffekt i framtidige forskningsprotokoller. Vi vil også få innsikt i om informasjon innsamlet ved innkomst kan gjøre klinikken i stand til å skreddersy oppfølging for pasientene. For pasienter med flere risikofaktorer for frafall kan man øke tiltak som er støttende. Dette har en del etiske aspekter som må tas hensyn til, for eksempel må det ikke brukes for å nekte enkelte pasienter med høy risiko for frafall tannlegebehandling. Den skal brukes som et arbeidsverktøy for å få pasienter gjennom tannbehandling. Totalt sett vil denne studien gjøre oss i stand til å vurdere om det er grunnlag for å implementere gratis tannhelsetjeneste som en del av behandlingstilbudet ved innleggelse til rusbehandling eller om en slik beslutning vil kreve større randomiserte studier.

### Utlysningsrelevans

Forskning innen tverrfaglig spesialisert behandling av rusavhengighet (TSB) er et prioritert område i Helse Nord sin Strategi for forskning og innovasjon i Helse Nord 2016-2020. Rusfri uten tannverk (RUST) er et tverrfaglig klinisk prosjekt der målsetningen er å få erfaring med og vurdere implementering av tannbehandling som en del av tilbudet til pasienter innlagt ved Russeksjon UNN Narvik. UNN Narvik har liten aktiv forskningsaktivitet og dette prosjektet er det første forskningsprosjektet ved Russeksjon UNN Narvik.

## Bakgrunn, kunnskapsstatus og forventet nytte

Allerede i Stortingsmelding 35 (2006-2007) «Tilgjengelighet, kompetanse og sosial utjevning - Framtidas tannhelsetjenester» blir rusavhengige trukket frem som en gruppe med store tannhelseproblemer. Stortingsmeldingen vektlegger viktigheten av reduksjon av sosiale ulikheter i tannhelse og har som målsetning å gi gratis tannhelsetjeneste til utsatte grupper 1.

Nå, mer enn 10 år senere, er mange rusavhengige fremdeles uten rettigheter til gratis tannhelsetjeneste. I sin kronikk i Tidsskrift for norske legeforening skriver Tordis Høifødt og medforfattere2: Som helsetjeneste må vi derfor sørge for at tannhelsen undersøkes og følges opp på linje med annen somatisk helse. I tillegg må lovverket justeres slik at de formulerte rettighetene tydeliggjøres, og det må klart og tydelig sikres at nødvendig tannbehandling faktisk gis vederlagsfritt til pasienter med alvorlige psykiske lidelser.

Både rusavhengige og tidligere rusavhengige opplever at dårlig tannhelse bidrar til mye tannpine, stigma og flere vanskeligheter i dagliglivet.

Det er sannsynlig at dårlig tannhelse med tilhørende smerteproblematikk, opptar pasientens kognitive kapasitet og hemmer annen behandlingstilnærming. Hvis et tilbud om tannhelsetjeneste som en integrert del av avhengighetsbehandlingen kan fungere som en «gulrot» for å søke seg til og møte opp til behandling, kan det også øke compliance under behandlingen fordi når dårlige tenner repareres blir pasienten kvitt sine tannsmerter.

Hvor tilgjengelig for behandling er en person som har tannsmerter og dårlig selvfølelse på grunn av manglende og råtnende tenner? Hvem vil ansette en person der smilet avslører råtne tannstubber?

## Dagens situasion ved UNN Russeksion Narvik

I dag har kun pasienter som er innlagt ved en avrusningsenhet i over tre måneder rett til gratis tannhelsehjelp3. Ved UNN Russeksjon Narvik er de fleste pasienter innlagt for en kortere periode enn tre måneder. Pasienter i LAR har tilgang til tannbehandling i den offentlige tannhelsetjeneste. Pasienter med tilbud fra kommunal hjemmetjeneste har fri tannhelsetjeneste. For begge grupper er erfaringen at de ikke har benyttet seg av sine rettigheter.

Om pasientene søker NAV om tilskudd til tannbehandling etter at de ankommer Russeksjon UNN Narvik vil søknaden sjelden være ferdig vurdert før behandlingsoppholdet er fullført. Hvis søknaden innvilges mens pasienten er innlagt, vil ventetiden til tannlegetime i den offentlige tannhelsetjenesten oftest være så lang at de ikke kan /får benyttet tilbudet under oppholdet.

Ved opphold under tre måneder vil kun akutte og nyoppståtte tannplager/smerter dekkes av klinikken eller spesialisthelsetjenesten med et maksimalbeløp på 1500 kr per tannbehandling. Fordi tannbevarende behandling er kostbart utføres det som oftest tannekstraksjoner, noe som ofte gir et lite tilfredsstillende funksjonelt og kosmetisk resultat.

Prosjekt RUST er relevant fordi prosjektet søker å øke vår kunnskap om ulike sider av om gratis tannhelsetjeneste bør implementeres som en del av behandlingstilbudet for alle som legges inn til rus/avhengighetsbehandling. Dette er kunnskap som er nyttig både for den enkelte pasient og for helsetjenesten som helhet.

Prosjekt RUST er også i tråd med visjonen som ble laget da man begynte planleggingen av Nye UNN Narvik: ..... "å utvikle en moderne helsetjeneste i Troms og Ofoten (TO) innenfor samhandlingsreformens prinsipper og rammevilkår, som kan være et "utstillingsvindu" og modell for andre regioner 4.

Arbeidet med å realisere sykehuset er nå i full gang og vi vil være i fortløpende kontakt med prosjektgruppene som jobber med planleggingen av det nye sykehuset, og jobbe for at et fullverdig tannlegekontor med tannlege og hjelpepersonell blir realisert til det beste for alle pasienter. Flere av prosjektgruppens medlemmer er med på planleggingen av det nye sykehuset.

Helsedirektoratets «Tannhelse – pakkeforløp for psykisk helse og rus»s tydeliggjør at rusbrukere er en befolkningsgruppe som bør prioriteres innen tannhelsetjenesten. Vi tenker derfor at tiden er moden for å høste erfaringer og studere gratis tannhelsetjeneste som en del av behandlingstilbudet ved UNN Russeksjon Narvik.

Nasjonale og internasjonale tall for rusbehandling viser at omkring halvparten av pasientene avslutter behandlingen før planlagt tidspunkt<sub>6,7</sub>.

Tabell 1. Drop-out fra TSB ved UNN 2014.

| | Utvalg | Andel |
|--------------------------------|--------|-------|
| Pasienthenvisninger | 414 | 100 % |
| Ikke møtt | 117 | 28 % |
| Møtte til behandling | 297 | 72 % |
| Avbrøt behandling | 98 | 33 % |
| Ikke møtt/avbrutt behandling | 214 | 52 % |
| Møtt og gjennomført behandling | 199 | 67 % |

Kilde: Kvaal B et al (2016)



# Tverrfaglig spesialisert behandling av ruslidelser (TSB)

Andelen som gjennomfører behandling varierer med institusjonstype? Ved tverrfaglig spesialisert behandling for rusmiddelavhengighet ved UNN (TSB UNN) gjennomførte 48% av de som ble henvist behandlingen (Intention to Treat), dette tilsvarer at 67% av de som møtte opp til behandling (Per Protokoll). Kvaliteten på rapporterte tall gjør at tallene for frafall er usikre og bør tolkes med forsiktighets

## Tannverk, tannstatus og tannbehandling blant rusmisbrukere

Det er godt dokumentert at forekomsten av dårlig tannstatus blant rusmisbrukere er høy 9–13, samtidig som dette er en pasientgruppe som i mindre grad enn befolkningen generelt oppsøker tannlege14,15. Dårlig tannhelse reduserer oral helserelatert livskvalitet målt med «Oral Health Impact Profile» også hos personer med rusproblmer16.

Det kan være mange grunner til at rusavhengige unngår å oppsøke tannlege: tiltaksløshet, rusbruk, fravær av smerter på grunn av rusbruk, tannlegeskrekk og manglende betalingsevne. Til tross for en høy forekomst av tannlegeskrekk uttrykker de fleste et ønske om tannbehandling under innleggelsen. Dette stemmer godt med andres erfaringer<sub>12</sub>.

Det er sannsynlig at dårlig tannstatus hos rusmisbrukere bidrar til udiagnostisert smerteproblematikk. Under behandling for rusavhengighet kan dårlig tannstatus øke risikoen for tannpine, dette kan igjen bidra til lavere motivasjon for rusfrihet. I en undersøkelse om tannhelse blant injiserende heroinmisbrukere i Oslo, oppga mer enn 35% tannsmerter som årsak til siste tannlegebesøk. Flere av deltakerne i studien fortalte også at tannverk hadde fått dem til å ruse seg under avrusing13.

Rusreformen i 2004 resulterte i pålegg om tannhelsetilbud til rusmiddelavhengige i rehabilitering17. Gratis tannhelsetjeneste til rusbrukere er utprøvd både utenfor og innenfor

sykehus<sub>10,12,17–19</sub>. Man har bekreftet at tannstatus er dårlig, og at ønsket om tannbehandling er stort, men ikke alle klarer å fullføre tannbehandlingen<sub>12,17</sub>.

I 2006 startet sykehus-tannhelseprosjektet ved TAKO-senteret(?) på Lovisenberg Diakonale Sykehus hvor det ble gitt midler for tannbehandling til pasienter med rusavhengighet og psykiatridiagnose 10. TAKO-senteret på Lovisenberg Diakonale Sykehus har gratis tannhelsetjeneste som en fast del av behandlingstilbudet ved sykehuset. Alle pasientene uttrykte tilfredshet med behandlingen, følte de fikk bedre tyggefunksjon, et mer akseptabelt smil og dermed større mulighet til fremtidig jobb og sosialt liv.

Ved Psykisk helse- og rusklinikken på UNN Tromsø har det lenge vært et tilbud om tannbehandling i samarbeid med Tromsø fylkeskommune19. Men for de fleste som legges inn til rus/avhengighetsbehandling der varigheten er under tre måneder finnes det ikke et slikt integrert tilbud.

Tannbehandling er et prioritert tiltak når pasienter stabiliseres i Legemiddel Assistert Rehabilitering (LAR), men dette forutsetter initialt tilstrekkelig compliance for gjennomføring av avrusning og stabilisering. For personer som er under rehabilitering for rusrelaterte problemer, og for personer som benytter seg av lavterskeltilbud for rusmisbrukere finnes følgende særskilte ordninger20:

- Fri behandling til rusmiddelmisbrukere som har vedtak etter Sosialtjenestelovens § 4-2 pkt a-d jfr § 4-3; de som ikke kan dra omsorg for selg selv, eller som er helt avhengig av praktisk eller personlig hjelp for å greie dagliglivets gjøremål, har krav på hjelp etter § 4-221. Dette forutsetter at pasientene mottar de nevnte tjenester i sammenhengende 3 måneder eller mer22.
- Noen tannhelsetjenester i lavterskel-helsetiltak for rusavhengige tilbyr fri tannlegebehandling.
- Fri tannbehandling til personer som mottar LAR.

Personer med rusproblemer kan søke NAV om Stønad til tannbehandling ved manglende evne til egenomsorg ved varig sykdom eller varig nedsatt funksjonsevne etter Lov om Folketrygd23 eller om stønad til tannbehandling ifølge Lov om sosiale tjenester grunnet økonomiske problemer24. Søknadsprosessen kan være tungvinn med behov for tilstrekkelig dokumentasjon og tidvis lang vurderingstid.

# Forventet nytte for pasienter

Ved å inkludere tannbehandling som en del av behandlingstilbudet for personer innlagt ved rusklinikker vil pasientene som mottar tilbudet oppnå bedre tannstatus, bedre egenopplevd tannhelse, bedre selvfølelse på grunn av mestring av tannlegeangst og et smil med sunne tenner. Vi tenker at dette øker sannsynligheten for at de klarer å nyttiggjøre tilbudene ved rusbehandlingen.

Om en pasient ikke klarer å gjennomføre hele tannhandlingen ved sitt opphold ved rusklinikken vil bedret tannhelse likevel kunne bidra til mindre smerter og høyere motivasjon til å oppsøke tannlege. Et tilbud om tannbehandling som en del av behandlingstilbudet vil kunne motivere personer med rusproblemer til å søke opphold ved rusklinikker som har dette tilbudet.

Som nevnt viser studier at omkring halvparten av de som starter rus/avhengighetsbehandling dropper ut før de er ferdigbehandlet<sub>6,7</sub>. Dette er en belastning både for den enkelte rusmisbruker som opplever det å mislykkes og for samfunnet som investerer i behandling som ikke gir de forventede resultatene. Hvis gratis tannbehandling reduserer drop-out og reinnleggelser vil dette føre til reduksjon i ventetid og bedre kapasitetsutnyttelse, gi bedre utnyttelse av de ansatte og dermed effektivisere driften. Selv med en ganske liten økning i gjennomføring og rusfrihet etter opphold, vil et slikt tilbud på landsbasis kunne ha stor betydning.

### Hvordan kan kunnskap fra studien tas i bruk i tjenesten

Basert på resultatene og erfaringene vil vi spre kunnskapen som genereres i prosjektet til viktige målgrupper og interessegrupper. Vi vil i løpet av studien samle erfaringer med tilbudet med tanke på om det er hensiktsmessig å jobbe videre for å implementere gratis tannhelsetjeneste som en del av det eksisterende behandlingstilbudet til rusavhengige eller om det trengs mere kunnskap før en slik implementering kan finne sted.

Hvis prosjektet lykkes og vi vurderer resultatene dithen at tilbud om gratis tannhelsetjeneste lar seg implementere i det eksisterende behandlingstilbudet, at de fleste som tar imot tilbud om tannbehandling er fornøyde og gjennomfører tannbehandlingen og at tannbehandlingen bidrar til bedret tannhelse, vil en naturlig konsekvens være en utvidelse av prosjekt RUST til andre institusjoner i Helse Nord. I så tilfelle vil det kreve en prioritering/omprioritering eller bevilgning av friske midler, tannhelsetjeneste er ikke gratis.

## Problemstillinger, hypoteser og metodevalg

## Drop-out fra behandling

Ideelt sett burde det gjennomføres randomiserte studier for å undersøke om gratis tannhelsetjeneste bidrar til redusert drop-out fra rus/avhengighetsbehandling, men før man vurderer å gjøre en randomisert studie er pilot/feasibilitystudie nødvendig for å vurdere om frafall fra både rus- og tannbehandlingen vil korrumpere RCT designet. En enkel styrkeberegning viser at det kreves at nærmere 800 pasienter inkluderes i en RCT for å vise reduksjon i drop-out fra 50% til 40%. I tillegg må det tas hensyn til at mange ikke klarer å gjennomføre tannbehandlingen, dette gir ulikt frafall av deltakere avhengig av om de er i kontroll eller intervensjonsgruppe og resulterer i «attrition bias/selection bias = frafallsskjevhet». Attrition bias er en trussel mot validiteten og generaliserbarheten av RCTer25.

## Gjennomføring av tannbehandling

Vår arbeidshypotese er at dårlig tannstatus med kronisk smerteproblematikk vanskeliggjør avrusning og stabilisering under døgnopphold under rus/avhengighetsbehandling. Det er naturlig å tenke at tidligere rusing har dempet tannsmertene og slik bidrar avrusning til å forsterke en ond sirkel med oppblussing av tannsmerter, ytterligere russug, dårlig compliance til avrusningsbehandling og i ytterste konsekvens drop-out (se figur).



Den norske retrospektive studien til Helvig og medarbeidere viste at mer enn 40% av rusmisbrukerne i studien ikke klarte å gjennomføre tannbehandling. Deltakerne i studien var rusmiddelavhengige under substitusjonsbehandling (LAR), rusmiddelavhengige som mottok kommunale hjelpetiltak, rusmiddelavhengige som oppholdt seg i institusjon i mer enn tre måneder og rusmiddelavhengige med psykiske og rusrelaterte problemer.

Studiepopulasjonen til Helvig og medarbeidere er ikke direkte sammenlignbare med de pasientene vi planlegger å inkludere ved UNN Russeksjon Narvik, og det er umulig å gjennomføre en RCT før man vet mer om frafall fra tannbehandling og får kunnskap om hvordan man kan øke andelen som gjennomfører tannbehandlingen for eksempel gjennom feasibility/pilotstudier.

Vi har derfor valgt å i denne omgang gjennomføre en ikke randomisert, intervensjonsstudie uten kontrollgruppe der intervensjonen er tilbud om tannbehandling og primært endepunkt er andel som gjennomfører denne. Studien vil inkludere 40-50 pasienter innlagt til rus/avhengighetsbehandling ved Russeksjon UNN Narvik. Studien er underdimensjonert med hensyn på primært endepunkt og den mangler kontrollgruppe. Vår overordnede målsetning er derfor å gjøre kvalitative vurderinger av kvantitativt innsamlede resultater.

Ut fra de funnene og erfaringene vi gjør i løpet av studien vil vi vurdere om en fremtidig studie kan/bør gjennomføres, og i så tilfelle hvordan26. Ut fra definisjonen på pilot/feasibilitystudier faller vårt randomiserte design uten kontrollgruppe inn under kategorien feasibilitystudie og vi har valgt å søke om midler for ett år slik at vi kan gjøre datainnsamlingen.

Primær målsetning for vår studie er å undersøke gjennomføringsgraden av tannbehandling i løpet av behandlingsperioden med vektlegging på assosiasjoner som øker sannsynlighet for gjennomføring og assosiasjoner som reduserer sannsynlighet for gjennomføring. Vi har ikke styrke til å gjøre avanserte korrelasjonsanalyser, men vi kan ved hjelp av deskriptive statistikk og enkle korrelasjoner gjøre kvalitative vurderinger av ulike statistiske sammenhenger og ut fra dette vurdere hva som er en hensiktsmessig fortsettelse.

I tillegg vil vi kartlegge hvilke assosiasjoner som øker sannsynlighet for gjennomføring av behandling. På basis av denne informasjonen vil vi modellere risiko for frafall fra tannbehandling. Vi vil så langt det er mulig innenfor de rammene til en ikke randomisert intervensjonsstudie kartlegge suksess- og fiaskofaktorer etterhvert som vi erfarer dem og vil i den grad det er mulig sette inn tiltak som øker sannsynlighet for suksess. Dette er så vidt vi vet ikke gjort tidligere i en populasjon av pasienter innlagt til rus/avhengighetsbehandling i en institusjon.

Utover disse to kvantitative målsettingene vil det utforskes om parallell tannbehandling har innvirkning på utbytte av rusbehandlingen, eller om det kan virke forstyrrende for gjennomføring. Videre søker studien å:

- ⇒ Vurdere om tannhelsetjeneste lar seg implementere som en del av det eksisterende behandlingstilbudet uten at det går utover annen behandling.
- ⇒ Beregne drop-out fra rus/avhengighetsbehandlingen for de som gjennomfører og de som ikke gjennomfører tannbehandlingen
- ⇒ Beregne faktiske behov for og kostnader ved tannbehandling
- ⇒ Vurdere om resultatene sammen med eksisterende kunnskap på feltet samlet er nok for å implementere gratis tannhelsetjeneste som en del av behandlingstilbudet ved rusproblemer.

# Gjennomføring av prosjektet

I forkant av prosjektperioden vil prosjektgruppen ha flere informasjonsmøter med ansatte i avdelingen der prosjektet presenteres skriftlig og muntlig. For å lykkes er vi helt avhengige av at de ansatte sitt samarbeid. Vi vil oppfordre de ansatte til å komme med innspill til forbedringer og gi uttrykk for skepsis som for eksempel til om det er mulig å presse flere tilbud inn i behandlingen. Før prosjektet kan gjennomføres er det nødvendig at ansatte er innforstått med hva som forventes av dem og hvordan vi sammen kan bidra til at gjennomføringen av prosjektet lykkes.

I tillegg til informasjonsmøter med ansatte vil vi før, under og etter studien gjennomføre spørreskjema- intervjuundersøkelse blant seksjonens personell med fokus hvordan prosjektet påvirker deres hverdag, kontakt/avtaler med pasientene og positive og negative sider ved implementering av gratis tannhelsetjeneste som en del av behandlingstilbudet ved UNN Russeksjon Narvik.

Sammen med innleggelsesbrevet fra UNN Russeksjon Narvik vil det følge et informasjonsbrev om prosjekt RUST. Pasientene vil få informasjon om prosjektet og forespørsel om å delta når de starter sin rus/avhengighetsbehandling ved døgnavdelingen. Svar på forespørsel om deltakelse vil ikke bli innhentet i en konsultasjons- eller behandlingssituasjon og vi vil ikke avkreve et aktivt nei-svar hvis en person ikke ønsker å delta. For å forhindre at forskningsdeltakeren føler seg presset til delta vil det informerte samtykket innhentes av en person som forskningsdeltakeren ikke har et avhengighetsforhold til, jf. helseforskningsloven § 13. Vi vil gi pasientene betenkningstid slik at de kan rådføre seg med andre før de avgjør om de ønsker å delta. For å sikre at deltakerne kan levere inn

samtykke på eget initiativ vil det bli satt opp låste postkasser der de som ønsker å delta kan legge samtykke.

Alle som ønsker å delta i studien tilbys tannlegetime så snart de er klare for dette. Tannlege Magnus Børseth vil vurdere behov for *nødvendig* tannbehandling. Tannbehandlingen vil bli utført mens pasienten er under rus/avhengighetsbehandling ved Russeksjon Narvik. Alle som deltar i intervensjonen vil i tillegg til klinisk tannundersøkelse bli bedt om å svare på noen spørsmål ved inklusjon i studien og etter avsluttet tannbehandling. De som ønsker hjelp til å fylle ut spørreskjema vil få dette. Deltakerne vil kunne ta kontakt med prosjektmedarbeiderne ved behov og få informasjon, støtte og hjelp. Hver deltaker er med i studien i den tiden han/hun er til behandling ved seksjonen og hvis det er praktisk mulig vil de få gjort ferdig planlagt tannbehandling etter de er ferdig med sin behandling ved Russeksjon UNN Narvik. All tannbehandling avsluttes om pasienten avbryter sin rus/avhengighetsbehandling ved Russeksjon Narvik (drop-out).

Vi vil avholde informasjonsmøter på UNN Russeksjon Narvik og informere om hvordan studien utvikler seg. Alle som er innlagt ved russeksjonen vil bli oppfordret til å gi tilbakemelding på hvordan studien påvirker deres hverdag.

Det vil bli satt opp låste postkasser der ansatte og innlagte ved UNN Russeksjon Narvik anonymt kan meddele prosjektgruppen sine meninger.

En del informasjon vil analyseres fortløpende for om mulig tilpasse studien innsigelser og gjøre forbedringer i logistikken omkring deltakerne.

Psykolog Patrik Nilsen vil foreta de kliniskpsykologiske undersøkelsene av deltakerne. Dette er rutineundersøkelser alle som legges inn ved russeksjonen gjennomgår.

Innsamlingen av data avsluttes når 100 deltakere har gjennomført behandingsoppholdet. Datamaterialet systematiseres og analyseres med utgangspunkt i primære og sekundære målsetninger. Studien avsluttes og data anonymiseres eller slettes tre år etter siste deltaker har gjennomført studien. Det vil ikke være noen kontrollgruppe i prosjektperioden, men vi vil kunne sammenlikne drop-out fra behandling med tidligere tall fra seksjonen og nasjonale tall.

#### **Brukermedvirkning**

Resultatene av dette forskningsprosjektet vil kunne brukes av helsetjenesten og helsebyråkratiet som helhet, den enkelte behandlingsenhet, forskergrupper/enkeltforskere og av personer som selv sliter med rus og avhengighetsproblematikk.

Esben Haldorsen er brukerrepresentant i prosjektgruppen. Han er representant for tidligere og nåværende rusbrukere og har selv vært pasient ved UNN Russeksjon Narvik, og har i perioden 2007-2010 hatt flere innleggelser der. Esben jobber til daglig som en av to ledere ved Exit Narvik, som er et brukerstyrt ettervernstilbud innenfor rus og psykisk helse. Exit Narvik driftes av brukerorganisasjonen Marborg og Esben har vært ansatt der siden 2012. Han har i perioden 2016-2018 vært nestleder i brukerutvalget ved UNN. Han brukes ofte som underviser både for pasienter og ansatte ved Russeksjon UNN Narvik. Han er medlem av prosjektgruppen for RUST. Han har vært med på utformingen av protokollen og kommet med innspill og forslag til forbedring. Esben Haldorsen og mange andre som har vært og er avhengige av rusmidler har erfaring med hvordan dårlig tannhelse bidrar til smerter og dårlig selvbilde og at gratis tannhelsetjeneste burde være en del av behandlingstilbudet til alle som sliter med rusproblemer.

## Samfunnsmessig relevans

Ifølge tall fra SSB27 hadde Tverrfaglig spesialisert rusbehandling 1896 døgnplasser med tilsammen 596.626 liggedager og i alt 17.730 utskrivinger i 2018. I snitt betyr dette litt i underkant av 34 liggedager pr utskriving. Totalt kostet Tverrfaglig spesialisert rusomsorg 5395 millioner kroner og hadde 4032 årsverk i 2018.

Vi mener at prosjekt RUST har stor samfunnsmessig relevans da det er med på å samle kunnskap om gratis tannhelsetjeneste kan bidra til å bedre rusbrukeres hverdag, øke motivasjon for behandling, redusere drop-out og gjøre flere i stand til å bidra i samfunnet. Selv små endringer i drop-out kan ha stor betydning for utnyttelsen av samfunnets ressurser.

### Innovasjon

Innføring av gratis tannhelsetjeneste som en integrert del av behandlingstilbudet for rusmisbrukere kan ses på som en tjenesteinnovasjon som vil bedre behandlingen av denne pasientgruppen.

## Miljøkonsekvenser

Vi kan ikke se at prosjektet har miljøkonsekvenser utover det som finner sted ved all (ordinær) tannbehandling.

#### Etikk

Rusbrukere er en sårbar gruppe og det må tas særlige hensyn til den enkelte deltakers behov. Vi vil være lydhøre overfor innspill fra deltakerne og i den grad det er mulig tilrettelegge for at hver enkelt deltaker føler seg ivaretatt mens studien pågår.

Det kan stilles spørsmålstegn ved at ektefellene Katrine og Magnus Flaaten Børseth begge er med i prosjektgruppen. Forklaringen på dette er at Magnus Flaatten Børseth i 2017 kontaktet Andreas Holund med spørsmål om det kunne være aktuelt å starte opp et prosjekt innen tannhelse hos rusmisbrukere. Det viste seg da at Andreas Holund alt hadde tatt opp emnet med flere lokale politikere, og han tok raskt "tenning" på ideen om å starte et samarbeid. Tanken var å få en bedre flyt innen tannbehandling hos rusmisbrukere, og helst at dette kunne bli en integrert del av behandlingen ved UNN Russeksjon Narvik. Katrine Flaatten Børseth var på dette tidspunktet tilknyttet UNN Russeksjon Narvik og det var naturlig at hun ble med i prosjektgruppen. Hun jobber nå som LIS II ved seksjonen.

De personene i prosjektgruppen som har daglig kontakt med deltakerne er alle ansatt ved UNN Russeksjon Narvik. Dette kan medføre at noen føler seg presset til å delta på studien, men vi vil i rekrutteringen ta hensyn til dette.

All informasjon som samles vil bli lagret sikkert på UNN sin forskningsserver. Hver deltaker vil få et løpenummer. Koblingsnøkkel mellom ID og løpenummer vil bli oppbevart på papir og være nedlåst.

Søknaden er vurdert av REK som en helsefaglig studie der funnene i studien indirekte vil kunne gi en helsemessig gevinst, men studien faller ikke inn under definisjonen av de prosjekt som skal vurderes etter helseforskningsloven (se vedlegg fra REK).

Søknad om godkjenning av prosjektet er sendt Personvernombud ved UNN. Det skal ikke samles inn biologisk materiale. Prosjektet starter ikke før godkjenning foreligger. Studien vil bli registrert i ClinicalTrials.gov før oppstart.

#### **Uheldige hendelse**

Uheldige hendelser vil bli dokumentert.

#### Kommunikasion og formidling

Resultatene fra studien vil bli publisert i et fagfellevurdert tidsskrift. Vi tenker at enten Tidsskrift for den norske Legeforening eller Norsk Tannlegeforening Tidsskrift er tidsskrifter der vi når flest mottakere som vil kunne ha nytte av resultatene fra studien. I tillegg vil medlemmer av prosjektgruppen holde foredrag og skrive innlegg i media om prosjektet.

### Søkermiljøet kompetanse

Gjennom sitt mangeårige arbeid som kliniker ved UNN Russeksjon Narvik har seksjonsoverlege Andreas Holund opplevd at svært mange pasienter miste motivasjon for rusbehandling med økende tannsmerter i forbindelse med avrusning. Siden få av pasientene ved seksjonen tilfredsstiller kravene til gratis tannbehandling eller av ulike årsaker ikke klarer å benytte seg av tilbudet hvis de tilfredsstiller lovverket utviklet han idéen om å teste ut gratis tannbehandling som en integrert del av behandlingstilbudet ved seksjonen. UNN Russeksjon Narvik mangler forskning og forskningskompetanse og han ønsket derfor å gjennomføre prosjektet som en klinisk intervensjonsstudie slik at man kunne samle og dokumentere erfaringene fra prosjektet og bruke disse for å evaluere om gratis tannbehandling kan være en nyttig del av behandlingen.

Prosjektleder Merethe Kumle er lege og epidemiolog og har erfaring med forskningsdesign og metode. Postdoktor og lege Terje Holmlund har gode statistiske metodekunnskaper og erfaring med statistisk bearbeiding av data. De vil begge ta aktivt del i gjennomføringen av prosjektet.

Psykolog Patrik Nilsen er ansvarlig for utvelgelse av spørreskjema. Han vil administrere innsamling av data og følge opp deltakerne under oppholdet. Lege Katrine Flaatten Børseth arbeider som Lege i spesialisering ved seksjonen, hun vil samle inn spørreskjema og intervjudata og vil gjennom prosjektet få erfaring med bearbeiding av data. Fagutviklersykepleier Stian Anthonsen vil ha det daglige ansvaret for innsamling av spørreskjema og hjelpe de av deltakerne som har spørsmål til studien eller som trenger hjelp til utfylling av skjema.

Tannlege Magnus Børseth vil undersøke deltakernes tenner og munnhule. Legge en individuell behandlingsplan for nødvendig tannbehandling og ha ansvaret for denne, Han vil samle inn tannbehandlingsdata i studien.

Esben Haldorsen er brukermedvirker. Han har selv vært rusmisbruker og har erfaring med hvordan dårlig tannstatus påvirker dagliglivet. Esben har vært aktivt med i utformingen av prosjektet og protokollen. Han vil være en viktig støttespiller for deltakerne i studien.

#### **Avslutning**

Flere av prosjektmedarbeiderne i dette prosjektet arbeider innen rus- og psykiatri, og de opplever nesten daglig at pasienter forteller om tannrelaterte plager som bidrar til å redusere oppmerksomheten om rus/avhengighetsbehandlingen når den smertedempende effekten av rusmidlene forsvinner.

Som vi har vist er dokumentasjonen for at tannbehandling bedrer tannhelse og oral helserelatert livskvalitet hos rusmisbrukere solid. Det samme er dokumentasjonen av at rusmisbrukere ønsker tannbehandling, men at de av ulike årsaker ikke klarer å gjennomføre denne på eget initiativ. Vi tenker derfor at dette prosjektets hovedoppgave er å knytte sammen kunnskap innhentet gjennom RUST med eksisterende kunnskap i håp om å bidra til at gratis tannhelsetjeneste implementeres som del av behandlingstilbudet til alle rusmisbrukere mens de er innlagt til behandling.

#### Referanser

- 1. Helse-og-omsorgsdepartementet. St.meld. nr. 35 (2006-2007). Tilgjengelighet, kompetanse og sosial utjevning Framtidas tannhelsetjenester. (2007).
- 2. Høifødt, T. S., Lund-Stenvold, E. & Høye, A. Ikke glem tennene. *Tidsskr. Den Nor. legeforening* (2018) doi:10.4045/tidsskr.18.0581.
- 3. Røynesdal, K. & Lundemo, H. *Utvidet fykleskommunalt tannhelsetilbud i 2006. Helse- og omsorgsdepartementet* https://www.regjeringen.no/globalassets/upload/kilde/hod/rus/2006/0003/ddd/pdfv/272988-rundskriv i-2 2006.pdf (2006).
- 4. Myrbostad, A. & Lauvsnes, M. *Konseptrapport UNN Narvik*. https://unn.no/Documents/Om-oss/Byggeprosjekter/Nye UNN Narvik/Konseptrapport nye unn narvik 251010.pdf (2010).
- 5. Helsedirektoratet. Tannhelse pakkeforløp for psykisk helse og rus. Ivaretakelse av somatisk helse og levevaner ved psykiske lidelser og/eller rusmiddelproblemer (gjelder fra 1. januar 2019). (2018) doi:10.9.2018.
- 6. Brorson, H. H., Ajo Arnevik, E., Rand-Hendriksen, K. & Duckert, F. Drop-out from addiction treatment: A systematic review of risk factors. *Clinical Psychology Review* vol. 33 1010–1024 (2013).
- 7. Kvaal, B., Øiern, T. & Harwiss, H. L. *Hindre drop-out fra rusbehandling*. https://oslo-universitetssykehus.no/seksjon/nasjonal-kompetansetjeneste-for-tverrfaglig-spesialisert-rusbehandling-tsb/Documents/Skriftserie web print.pdf (2016).
- 8. Helsedirektoratet. Avbrudd i tverrfaglig spesialisert rusbehandling. https://www.helsedirektoratet.no/statistikk/statistikk/kvalitetsindikatorer/rusbehandling/avbrudd-i-tverrfaglig-spesialisert-rusbehandling.
- 9. Baghaie, H., Kisely, S., Forbes, M., Sawyer, E. & Siskind, D. J. A systematic review and meta-analysis of the association between poor oral health and substance abuse. *Addiction* (2017) doi:10.1111/add.13754.
- 10. Haugbo, H. O., Storhaug, K. & Willumsen, T. Rusavhengighet, psykiatri og oral helse. Rapport fra et sykehusprosjekt i Oslo Den norske tannlegeforenings Tidende. *Nor Tann. Tid* 13, 912- (2010).
- 11. Karlsen, L. S., Wang, N. J., Jansson, H. & Arnsteinsson, V. Tannhelse og oral helserelatert livskvalitet hos et utvalg rusmiddelmisbrukere i Norge. *Nor Tann. Tid* **127**, 316–21 (2017).
- 12. Karlsen, L. S. & Toven, H. V. *Tannbehandlingstilbud til og tannhelseforhold hos rusmiddelmisbrukere og personer med kvalifiseringsstønad fra NAV*. https://helsedirektoratet.no/Documents/Tannhelse/Sluttrapport for utredningsoppdrag tannhelse og rus 2015.pdf (2015).
- 13. Vanberg K, Husby I, Stykket L, Young A & Willumsen T. Tannhelse blant et utvalg injiserende heroinmisbrukere i Oslo. *Nor Tann. Tid* **126**, 528–34 (2016).
- 14. Grytten, J., Skau, I. & Holst, D. Tannhelsetjenestetilbudet blant voksenbefolkningen i Norge Den norske tannlegeforenings Tidende. *Nor Tannlegeforen Tid* 276–83 http://www.tannlegetidende.no/i/2014/4/d2e1061 (2014).
- 15. Hustvedt, I. B., Lie, T., Emmerhof;, Håland, M. E., Barclay;, S. & Nesvåg, S. *Tjenestemottakere med rus-og psykiske helseproblemer i kommunene*. http://www.brukerplan.no/BrukerPlanÅrsrapport2017 Digital.pdf (2018).
- van Wijk, A. J., Molendijk, G. & Verrips, G. H. W. OHRQoL in a Sample of Alcohol and Drug Abusers. *Open Dent. J.* (2016) doi:10.2174/1874210601610010338.
- 17. Helvig, J. I., Jensdottir, T. & Storesund, T. Har gratis tannhelsetilbud til rusmiddelavhengige ført til forventet effekt? *Nor Tann. Tid* **127**, 774–80 (2017).
- 18. Helvig, J. I. Erfaringer fra fire års offentlig tannlegepraksis for rusmiddelavhengige i Stavanger. *Nor Tann. Tid* **121**, 234–6 (2011).
- 19. Helsedirektoratet. Evaluering av «Forsøksordning med orale helsetjenester organisert i tverrfaglig miljø ved sykehus. (2019).
- 20. Olsø, T. M. Rettigheter til fri tannbehandling NAPHA Nasjonalt kompetansesenter for psykisk helsearbeid. https://www.napha.no/content/14163/Rettigheter-til-fri-tannbehandling (2010).
- 21. Myhre, L. & Lossius, M. C. Ber om avklaring ift. tolkning av Lov om sosiale tjenester § 4-3, JF. § 4-2 C Støttekontakt | Helsetilsynet. https://www.helsetilsynet.no/regelverk/tolkningsuttalelser/helse-omsorgstjenester/ber-avklaring-ift-tolkning-lov-sosiale-tjenester-4-3-jf-4-2-c-stoettekontakt/ (2008).
- 22. Helse- og Omsorgsdepartementet. I-2/2006. Utvidet fylkeskommunalt tannhelsetilbud i 2006. 048101-250006 (2006).
- 23. Arbeids og sosialdepartementet. *Lov om folketrygd (folketrygdloven) Lovdata*. https://lovdata.no/dokument/NL/lov/1997-02-28-19/\*#\* (1997).
- 24. Arbeids og sosialdeparetementet. Lov om sosiale tjenester i arbeids- og velferdsforvaltningen (sosialtjenesteloven) Kapittel

  1. Lovens formål og virkeområde Lovdata. https://lovdata.no/dokument/NL/lov/2009-12-18131/KAPITTEL 1#KAPITTEL 1 (2009).
- 25. Mansournia, M. A., Higgins, J. P. T., Sterne, J. A. C. & Hernán, M. A. Biases in randomized trials. *Epidemiology* **28**, 54–59 (2017).
- 26. Eldridge, S. M. et al. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ 355, i5239 (2016).
- 27. SSB.no. Tverrfaglig spesialisert rusbehandling. *Spesialisthelsetjenesten SSB* https://www.ssb.no/helse/statistikker/speshelse/aar (2019).